CLINICAL TRIAL: NCT01498224
Title: ReSure Sealant Pivotal Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OTX-11-002
Record Dates: First submitted 2011-12-18; First posted 2011-12-23 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-02

CONDITIONS: Cataract Surgery Incision Leak
Keywords: Cataract surgery
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture (Active Comparator): Suture application
  Interventions: Procedure: Sutures
- ReSure Sealant (Experimental): Sealant application
  Interventions: Device: ReSure Sealant

INTERVENTIONS:
Device: ReSure Sealant — Comparison of ReSure Sealant to suture(s)
  Arms: ReSure Sealant
Procedure: Sutures
  Arms: Suture

SUMMARY:
This is a randomized multicenter study to evaluate the safety and effectiveness of ReSure Sealant compared to sutures for preventing incision leakage within the first 7 days of cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a cataract and is expected to undergo clear cornea cataract surgery with phacoemulsification and implantation of posterior chamber intraocular lens
* Subject must be 22 years of age or older

Exclusion Criteria:

* Any intraocular inflammation in study eye or presence of ocular pain in operative eye at preoperative assessment
* Previous corneal or retinal surgery or planned multiple procedures during cataract surgery.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes with any clear corneal incision/suture leakage as determined by positive Seidel test indicating fluid egress within first 7 days after surgery. | Days 1-28

SECONDARY OUTCOMES:
Foreign Body Sensation | Days 1-28
Best corrected visual acuity | Day 1
  Best corrected visual acuity worse than 20/40 at day 1
Best corrected visual acuity | Day 28
  Best corrected visual acuity worse than 20/40 at 28 days

OTHER OUTCOMES:
Presence of ReSure Sealant or suture(s) | Day 28
  Presence of ReSure Sealant or suture(s)at every follow-up visit
Presence of blue colorant in ReSure Sealant | Day 28
  Presence of blue colorant in ReSure Sealant at every follow-up visit
Device ease of use | Day 0
  Device ease of use during application
Corneal edema at 1 day | Day 1
  Corneal edema at 1 day (moderate to severe stromal edema)
Anterior chamber inflammation | Day 1
  Anterior chamber inflammation (defined as greater than or equal to grade 2+ anterior chamber cells) at day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Levenson Eye Associates, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data is available on FDA website for approved PMA P130004

REFERENCES:
- See also: Publications of study results — http://www.resuresealant.com